CLINICAL TRIAL: NCT00898417
Title: Development of a Serum Proteomic Classifier for the Prediction of Benefit From Bevacizumab in Combination With Carboplatin and Paclitaxel
Brief Title: Biomarker Study of Blood Samples From Patients With Non-Small Cell Lung Cancer Treated With Carboplatin and Paclitaxel With or Without Bevacizumab
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000592948; ECOG-E4599T2
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; recurrent non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung; bronchoalveolar cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Bevacizumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Biological: bevacizumab
Drug: carboplatin
Drug: paclitaxel
Genetic: proteomic profiling
Other: laboratory biomarker analysis
Other: matrix-assisted laser desorption/ionization time of flight mass spectrometry

SUMMARY:
RATIONALE: Studying samples of blood in the laboratory from patients undergoing treatment for non-small cell lung cancer may help doctors predict how patients will respond to treatment.

PURPOSE: This laboratory study is looking at proteomic patterns in stored blood samples from patients undergoing treatment for non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To develop a serum proteomic classifier using matrix-assisted laser-desorption/ionization time-of-flight mass spectrometry analysis of blood samples from patients with non-squamous cell non-small cell lung cancer to predict benefit, in terms of survival and time to progression, from treatment with bevacizumab in combination with carboplatin and paclitaxel.

Secondary

* To better quantitate candidate biomarkers by using more advanced mass spectrometric technologies, including multiple-reaction monitoring and heavy-labeled peptides.

OUTLINE: Previously collected pre-treatment samples of serum or plasma are randomly selected from patients enrolled on protocol ECOG-4599 (i.e., 60 from the bevacizumab arm and 30 from the control arm). Samples are analyzed by matrix-assisted laser-desorption/ionization time-of-flight mass spectrometry to identify patterns from protein spectra that correlate with patient survival.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Available serum and plasma samples from patients with previously untreated locally advanced, metastatic, or recurrent non-squamous cell non-small cell lung cancer
* Enrolled on clinical trial ECOG-4599

  * Treated with carboplatin and paclitaxel with or without bevacizumab

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples submitted for research from patients participating in E4599
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2008-03-14 (Actual); Primary Completion 2008-04-14 (Actual); Study Completion 2008-04-14 (Actual)

PRIMARY OUTCOMES:
Survival | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: David P. Carbone, MD, PhD, Study Chair — Vanderbilt-Ingram Cancer Center